CLINICAL TRIAL: NCT05986214
Title: Developing an Intervention to Optimize Virtual Care Adoption for COPD Management (CDA 21-187)
Brief Title: Developing an Intervention to Optimize Virtual Care Adoption for COPD Management
Acronym: VC-OPTIONS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 23-001; CDA 21-187 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Disease, Chronic Obstructive; Telemedicine; Text Messaging; Implementation Science; Community-Based Participatory Research
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: All patient participants will all be assigned to the VC-OPTIONS implementation strategy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VC-OPTIONS (Experimental): Participants will be enrolled in the Annie texting VC-OPTIONS protocol
  Interventions: Other: VC-OPTIONS

INTERVENTIONS:
Other: VC-OPTIONS — Participants will be enrolled in the Annie texting VC-OPTIONS protocol
  Other Names: Texting Intervention

SUMMARY:
VA is a leader in virtual care (VC), including the patient portal, mobile apps, and telehealth programs. VC has great utility for managing chronic conditions like chronic obstructive pulmonary disease (COPD). However, adoption of many VC services has been slow. Lack of awareness about these services is one of the most prominent patient- and healthcare team-facing barriers to adopting VC. This study will develop, refine, and pilot a stakeholder-informed multicomponent implementation strategy to support adoption of VC, referred to as VC-OPTIONS (Virtual Care for Chronic Obstructive Pulmonary Disease Adoption Support). This feasibility trial will pilot the VC-OPTIONS implementation strategy to assess feasibility and acceptability and gather preliminary effectiveness data to inform a larger hybrid effectiveness-implementation trial. The core component of VC-OPTIONS will be the provision of information via VA's Annie texting program to empower patients with knowledge about the array of VC services and how they can be used to support COPD management. It is hypothesized that this strategy will be acceptable and feasible. This work will improve patient and team awareness of and communication about VC services, and support patient access to VC services for COPD management.

DETAILED DESCRIPTION:
VA is a leader in virtual care (VC), including the patient portal, mobile apps, and telehealth programs. VC has great utility for managing chronic conditions like chronic obstructive pulmonary disease (COPD). However, adoption of many VC services has been slow. Lack of awareness about these services is one of the most prominent patient- and healthcare team-facing barriers to adopting VC. This study will develop, refine, and pilot a stakeholder-informed multicomponent implementation strategy to support adoption of VC, referred to as VC-OPTIONS (Virtual Care for Chronic Obstructive Pulmonary Disease Adoption Support). This single-arm pilot will assess the feasibility and acceptability of VC-OPTIONS, as well as engagement and preliminary effectiveness specific to VC adoption, such as change in patient awareness of VC services. The investigators hypothesize that developing educational content about VC that can be delivered via text messaging will be an effective way to empower Veterans with knowledge and support them in their decision to adopt VC if they are interested.

Setting and design.

This feasibility pilot will be conducted at the VA Bedford and/or Boston Healthcare Systems. This pilot study will use quantitative data to assess patient and team perceptions of feasibility and acceptability, and preliminary effectiveness of the intervention. VC-OPTIONS will include patient- and team-facing strategies. The core component will be the delivery of educational content about VC for COPD via Annie text messaging. Other patient- and healthcare team-facing strategies will be refined in prior, preparatory aims.

Patient level. 40 eligible and interested Veterans will be assigned to the core patient-facing implementation strategy, the Annie texting protocol. Preparatory work will shape final length of protocol, content, and frequency of messages. The texting protocol as currently envisioned will span 12 weeks (1 module [Appendix 5] with up to 5 messages per week, and 2 messages every 4 weeks that ask about behavioral intention). Participants will receive compensation for initial baseline assessments and additional compensation after completion of the follow-up assessments.

Team-level. Pre-implementation meetings with local clinical team stakeholders (e.g., leadership, clinical team members, local telehealth/connected care coordinators) will be held to discuss site-level needs and contextual factors. Potential team-facing strategy components, developed during preparatory aims, will be presented and discussed to reach consensus and finalize the team-facing strategy components that are tailored to the site-level needs and resources.

Data collection. Patient-level. Recruitment procedures will be evaluated to inform a subsequent larger trial by examining how many potential participants agreed to participate in the intervention (feasibility and acceptability), and documenting reasons Veterans declined to participate. Participants will complete a baseline survey in person or over the phone to gather participant characteristics, VC awareness, current use of VC, and intent to use VC. Using Annie's two-way texting feature and dashboard, objective data will be collected on participant engagement during the protocol (i.e., how frequently participants respond to the texts, which patients received which modules, and completion rates). Engagement will also be assessed via survey at the post-evaluation. After completion of the texting protocol and clinical visit, data will be obtained via survey on the feasibility and acceptability of the core implementation component using the Feasibility of Intervention, Acceptability of Intervention, and Intervention Appropriateness measures. Preliminary effectiveness data will be gathered via surveys and clinical chart review on participants' awareness of VC, intention to adopt one or more VC options, intention to discuss VC with their clinical team, occurrence of patient-team communication about VC, and impact on COPD management.

Team-level. Clinical team perceptions of feasibility and acceptability will be measured quantitatively, such as through a brief survey to clinical team members who were exposed to the implementation components (e.g., those who attended the educational meetings, those who participated in clinical visits with participants who were enrolled in the texting protocol). Engagement will be measured by examining attendance of educational meetings. Preliminary effectiveness outcomes data will also be collected, including survey and chart-review to identify occurrence of conversations with patients about VC services (anticipated primary outcome of future IIR) and referrals to the Virtual Health Resource Centers or telehealth services and surveys to evaluate awareness of VC services before/after strategy deployment.

Data analysis. Summary statistics will be used to examine measurements and assess for perceptions of feasibility, acceptability, and preliminary effectiveness of the implementation strategy. The strategy components (the texting protocol, recruitment, and data collection procedures) will further be refined based on what is learned. Inferential analyses (paired t-tests or Wilcoxon signed rank tests) will be used to estimate effect sizes of changes between pre/post timepoints within individual participant. This feasibility pilot is not intended or powered to detect statistically significant changes in outcomes. Additionally, this pilot with no prospective control arm cannot definitively ascertain whether VC-OPTIONS causes leads to changes in effectiveness. These preliminary analyses seek to inform the design and generate effect size estimates.

ELIGIBILITY:
Inclusion Criteria:

* VHA user
* US Veteran
* COPD diagnosis
* the ability to speak and understand English
* own a text-enabled phone

Exclusion Criteria:

* Prior participation in preparatory research for the development of the intervention

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 12 Weeks
  The feasibility of the core implementation component will be assessed with the Feasibility of Intervention Measure (FIM). This is a publicly available, psychometrically sound scale designed to be used in pilot studies as an indicator of implementation success. Participants will be asked to indicate the extent to which they agree with the following statements on a scale from 1 (completely disagree) to 5 (completely agree): I can see other Veterans receiving these messages; I was able to respond to the text messages; texting with Annie was easy; the amount of messages I received from Annie was just right.

SECONDARY OUTCOMES:
Acceptability | 12 Weeks
  The acceptability of the core implementation component will be assessed with the Acceptability of Intervention Measure (AIM). This is a publicly available, psychometrically sound scale designed to be used in pilot studies as an indicator of implementation success. Participants will be asked to indicate the extent to which they agree with the following statements on a scale from 1 (completely disagree) to 5 (completely agree): I approved of the text messages I received; the text messages I received were appealing to me; I liked receiving and responding to the text messages I received; I welcomed the text messages I received.
Appropriateness | 12 Weeks
  The appropriateness of the core implementation component will be assessed with the Intervention Appropriateness Measure (IAM). This is a publicly available, psychometrically sound scale designed to be used in pilot studies as an indicator of implementation success. Participants will be asked to indicate the extent to which they agree with the following statements on a scale from 1 (completely disagree) to 5 (completely agree): the text messages were fitting; the text messages were suitable, the text messages were applicable to me; the text messages were a good match with my COPD management needs.
Awareness of Virtual Care | 12 Weeks
  Change between baseline and 12 weeks in awareness of Virtual Care services will be assessed via survey, pre and post intervention, through the following question: which of the following VA services are you aware of?
Intention to Adopt Virtual Care | Baseline and 12 weeks
  Change between baseline and 12 weeks in awareness of Virtual Care services will be assessed via survey through the following question: which of the following VA services are you interested in trying out?
Intent to Communicate about Virtual Care | Baseline and 12 weeks
  Change between baseline and 12 weeks will assess intent to communicate about Virtual Care from baseline to post-intervention (12 weeks) through the following questions: how interested are you in discussing these different services with your healthcare team; and how prepared do you feel to discuss these different services with your healthcare team? Participants will indicate on a 4-point scale from "not very" to "very."
Impact of COPD Management | 12 weeks
  Participants will be asked to describe via free text any impacts participation in this study has had on how they use technology to manage their COPD. This will be qualitative data.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Robinson, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (2):
- United States (2):
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. Data will be used by the research team only to inform manuscripts and future grant submissions.